CLINICAL TRIAL: NCT01291836
Title: Acute Kidney Injury Neutrophil Gelatinase-Associated Lipocalin (N-GAL) Evaluation of Symptomatic Heart Failure Study (AKINESIS)
Brief Title: Acute Kidney Injury Neutrophil Gelatinase-Associated Lipocalin Evaluation of Symptomatic Heart Failure Study
Acronym: AKINESIS
Status: Completed | Type: Observational
Sponsor: Alere San Diego (Industry)
Collaborators: Abbott Diagnostics Division (Industry); Alere, Inc. (Industry)
Responsible Party: Sponsor
Organization: Abbott RDx Cardiometabolic (Other)
Other Study IDs: DDDP-09EE-081
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Acute Decompensated Heart Failure; Acute Kidney Injury
Keywords: Acute Kidney Injury (AKI); Acute Decompensated Heart Failure (ADHF); Neutrophil Gelatinase Associated Lipocalin (NGAL); biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Samples, Plasma Samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
AKINESIS is a clinical study to assess the utility of blood and urine NGAL tests in predicting worsening kidney function in patients who present with acute heart failure (AHF) and who are treated with diuretics. It is believed that rising NGAL levels in the blood and/or urine can predict acute kidney injury. It is also believed that patients who are admitted to the hospital with high NGAL levels in the blood/urine will have poorer outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age.
* Subjects must present to the hospital with one or more signs or symptoms of acute heart failure (AHF). Signs and symptoms include shortness of breath from walking, rales or crackles, galloping heart rhythm, jugular venous distension, trouble breathing at rest or when lying down, waking breathless at night, using more than 2 pillows to sleep, tiring easily, swelling of feet, ankles or legs, frequent coughing, a cough that produces mucous or blood-tinged sputum, or a dry cough when lying flat.
* Subjects must receive IV diuretics, or there must be an intent to treat with IV diuretics.
* Subjects must be willing and able to comply with all aspects of the protocol.
* Subjects must provide signed informed consent.

Exclusion Criteria:

* Subjects that present with symptoms consistent with acute coronary syndromes (AMI or UA) as the chief cause of the current episode of AHF.
* Subjects already on dialysis prior to enrollment or if dialysis initiation is already planned during the current hospital visit.
* Subjects that have had any major organ transplant (heart, lung, kidney, or liver).
* Subjects that have participated in a drug treatment study within the past 30 days or if they have already been enrolled as a subject in this study.
* Women who verbally report being pregnant at the time of screening and anyone belonging to a vulnerable population that is deemed inappropriate for inclusion into the study by the IRB/EC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled primarily from hospital emergency rooms located at various academic centers located throughout the USA and Europe.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maisel, MD, Principal Investigator — University of California, San Diego Medical Center/Veterans Affairs Medical Center, San Diego; Patrick Murray, MD, Principal Investigator — University College of Dublin School of Medicine and Medical Science/Mater Misericordiae University Hospital
Locations (13):
- United States (6):
  - University of California San Diego Medical Center, San Diego, California
  - San Diego Veterans Administration Hospital, San Diego, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - New York Methodist Hospital, Brooklyn, New York
  - Virginia Commonweath University Medical Center, Richmond, Virginia
- Athens University Hospital Attikon, Athens, Greece
- University Hospital Dublin, Dublin, Ireland
- Italy (2):
  - Clinica Mediterranea, Naples
  - Monasterio Foundation for Medical Research and Public Health, Pisa
- University of Groningen Medical Center, Groningen, GZ Groningen, Netherlands
- Hospital Clínico Universitario Valencia, Valencia, Spain
- Universitätsspital Basel, Basel, Petersgraben, Switzerland

REFERENCES:
- [Derived] Duff S, Wettersten N, Horiuchi Y, van Veldhuisen DJ, Raturi S, Irwin R, Cote JM, Maisel A, Ix JH, Murray PT. Absence of Kidney Tubular Injury in Patients With Acute Heart Failure With Acute Kidney Injury. Circ Heart Fail. 2024 Nov;17(11):e011751. doi: 10.1161/CIRCHEARTFAILURE.123.011751. Epub 2024 Oct 18. PMID 39421939
- [Derived] Maisel AS, Wettersten N, van Veldhuisen DJ, Mueller C, Filippatos G, Nowak R, Hogan C, Kontos MC, Cannon CM, Muller GA, Birkhahn R, Clopton P, Taub P, Vilke GM, McDonald K, Mahon N, Nunez J, Briguori C, Passino C, Murray PT. Neutrophil Gelatinase-Associated Lipocalin for Acute Kidney Injury During Acute Heart Failure Hospitalizations: The AKINESIS Study. J Am Coll Cardiol. 2016 Sep 27;68(13):1420-1431. doi: 10.1016/j.jacc.2016.06.055. PMID 27659464

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrollment Group: Subjects with sufficient data to be included in the analysis.
- Subjects Enrolled But Not Included in the Analysis.: Subjects that were consented and some study procedures completed but did not have required study procedures completed and subsequent data available for inclusion in the primary analysis.
Period: Overall Study
Arm/Group | Enrollment Group | Subjects Enrolled But Not Included in the Analysis.
Started | 930 | 71
Completed | 930 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ED presentation with symptoms of Heart Failure.
Groups:
- Enrollment Group-No Treatment Arms.: All subjects underwent the same protocol procedures no stratification.
Arm/Group | Enrollment Group-No Treatment Arms.
Number analyzed (Participants) | 930
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 344
  >=65 years | 586
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354
  Male | 576
Region of Enrollment [Number; unit: participants]
  Greece | 27
  Netherlands | 97
  United States | 587
  Ireland | 41
  Italy | 110
  Switzerland | 52
  Germany | 1
  Spain | 15

OUTCOME MEASURES:

1. Primary Outcome: Evaluating the Efficacy of the Triage NGAL Test as an Aid to Diagnosis of Acute Kidney Injury (AKI) in Patients Admitted to the Hospital With Symptoms of Acute Heart Failure.
Description: Efficacy determined by the evaluation of the area under the Receiver Operator Curve (ROC) generated from the study primary endpoint data. The units on both axes of the ROC curve are dimensionless proportions from 0 to 1.
Time Frame: First week of hospitalization.
Population: Participants were enrolled from patients presenting to the ED with signs and/or symptoms of Heart Failure. Subjects also had to meet specific operational requirements for the blood drawing time frame, per the protocol.
Measure: Number (95% Confidence Interval); unit: Probability classifying AKI from non-AKI
Groups:
- Enrollment Group: Subjects enrolled in the study and completing required procedures to be included in the primary analysis.
Arm/Group | Enrollment Group
Number analyzed (Participants) | 930
Probability classifying AKI from non-AKI | 0.658 [0.586 to 0.730]
Statistical Analysis 1: Comparison: Enrollment Group; Null Hypothesis: ROC AUC of 0.58; using a one-sided z-test at a significance level of 0.025. Efficacy determined by the evaluation of the area under the Receiver Operator Curve (ROC) generated from the study primary endpoint data. The units on both axes of the ROC curve are dimensionless proportions from 0 to 1; Test type: Superiority or Other; Area under Receiver-Operator Curve (ROC) = 0.658, 95% CI 2-sided [0.586 to 0.73]; Efficacy determined by the evaluation of the area under the Receiver Operator Curve (ROC) generated from the study primary endpoint data. The units on both axes of the ROC curve are dimensionless proportions from 0 to 1

2. Primary Outcome: Evaluating the Efficacy of the Triage NGAL Test as an Aid in Predicting Poorer Outcomes in Patients Admitted to the Hospital With Admitted With Symptoms of Acute Heart Failure.
Description: as for outcome 1
Time Frame: ~30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability classifying AKI from non-AKI
Groups:
- Enrollment Group: Subjects enrolled and completing the required study procedures for the primary analysis.
Arm/Group | Enrollment Group
Number analyzed (Participants) | 930
Probability classifying AKI from non-AKI | 0.650 [0.598 to 0.702]
Statistical Analysis 1: Comparison: Enrollment Group; Null Hypothesis: AUC ≤0.55, using a one-sided z-test at a significance level of 0.025. Efficacy determined by the evaluation of the area under the Receiver Operator Curve (ROC) generated from the study primary endpoint data. The units on both axes of the ROC curve are dimensionless proportions from 0 to 1; Test type: Superiority or Other; ROC AUC = 0.650, 95% CI 2-sided [0.598 to 0.702]; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: ~30 days.
Groups:
- Enrollment Group: Subjects enrolled in the study and completing study procedures required for the analysis.
- Non-participating Group: Subjects consented and/or enrolled in the study but not completing study procedures required for the analysis.
Arm/Group | Enrollment Group | Non-participating Group
Serious Adverse Events (participants affected / at risk) | 0/930 | 0/71
Other Adverse Events (participants affected / at risk) | 0/930 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other